CLINICAL TRIAL: NCT02019888
Title: Comprehensive Wide Bandwidth Test Battery of Auditory Function in Veterans
Brief Title: Wide Frequency Band Test of Hearing in Veterans
Acronym: CWTBAFV
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Father Flanagan's Boys' Home (Other)
Responsible Party: Sponsor
Other Study IDs: C1268-R
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Otosclerosis; Tympanic Membrane Perforation; Otitis Media With Effusion; Cholesteatoma
Keywords: Ear, Middle; Ear, Inner; Audiometry; Acoustic impedance tests
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Otosclerosis; Tympanic Membrane Perforation; Otitis Media with Effusion; Cholesteatoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Normal hearing adults: Adults between 20 and 79 years old with hearing at all audiometric frequencies between 250 and 8000 Hz at less than or equal to 25 dB HL
- Adults with sensory neural hearing loss: Adults between 20 and 79 years old with sensory neural hearing at one or more audiometric frequencies between 250 and 8000 Hz.
- Adults with middle ear disorders: Adults between 20 and 89 years old with middle ear disorders: tympanic membrane perforation, serous otitis media, cholesteatoma, otosclerosis, and unspecified middle ear disorders.

SUMMARY:
The accurate assessment of auditory status is critical for planning treatment for Veterans with hearing loss to include medical and audiological management. Current physiologic tests of auditory function in the standard clinical audiological test battery for Veterans have limited sensitivity in detecting some middle-ear disorders, and do not include a direct test of cochlear function. Recent studies have shown promise for new wide-bandwidth (WB) tests of absorbance for improved sensitivity in the assessment of middle-ear function including acoustic reflex testing. The addition of WB tests of cochlear function included in the WB test battery provides an opportunity to improve audiological diagnosis of a range of hearing disorders in Veterans. The automation provided by the WB test battery could provide additional benefits in reducing the duration of the evaluation, leaving more time for evaluation of test findings and counseling. Results from this study may lead to the improvement of audiological care for Veterans with hearing loss.

DETAILED DESCRIPTION:
The goal of this research is to evaluate a comprehensive test battery of new wide-bandwidth, i.e., wideband (WB), acoustical tests of auditory function in the differential diagnosis of middle ear, cochlear and neural pathologies in a population of Veterans. WB tests refer to ear canal tests using sound responses measured from 0.2 kilohertz (kHz) to frequencies as high as 8 kHz, a bandwidth that is critical for speech perception. There will be tests in the battery for middle-ear assessment using power absorption, cochlear assessment using otoacoustic emissions (OAEs) and the acoustic stapedius reflex (ASR) using middle ear power absorption. Results will be compared with a standard single-frequency clinical immittance test battery routinely used in the assessment of auditory function in Veterans. Aim 1 seeks to evaluate the accuracy of the WB test battery in the differential diagnosis of middle-ear pathology and related conductive hearing loss by comparing the sensitivity and specificity of the WB battery to the traditional immittance battery for the following disorders common in Veterans: tympanic membrane perforation, serous otitis media, cholesteatoma, and otosclerosis. Aim 2 seeks to modify a WB ASR test to provide automatic detection of the ASR threshold for comparison with the traditional single-frequency ASR threshold. Aim 3 seeks to validate the use of Transient-evoked otoacoustic emission (TEOAE) and spontaneous otoacoustic emissions (SOAEs)tests in Veterans to assess cochlear status, and evaluate their test performance in classifying ears with normal hearing and sensorineural hearing loss. Finally, Aim 4 seeks to compare the diagnostic accuracy of the full WB test battery with the full single-frequency admittance test battery to detect any type of hearing loss including sensorineural, conductive and mixed. The hypothesis is that the WB test battery is more accurate than the traditional immittance test battery in identifying ears with normal auditory status and ears with a range of risks for auditory pathology.

Methods:

Subjects- Human subjects will be recruited for this study who have had a hearing evaluation from the VA Audiology Service at the Portland VA Medical Center and the H. Quillen VA Medical Center. These subjects will respond to flyers or be contacted from an IRB-approved human subject volunteer registry. Additional details regarding recruitment and selection criteria may be found in the next sections of the protocol. The investigators will recruit approximately equal numbers of subjects, with a total of 640. Data will be acquired at the two sites from a total of 190 adult subjects with normal hearing and 180 adult subjects with sensorineural hearing loss. These subjects will be recruited from three age groups: 20-39 years, 40-59 years and 60-79 years for age comparisons of normative middle-ear data. Data will also be acquired at both sites from 250 adult subjects with middle-ear disorders and/or conductive hearing loss from ages 20-89 years. Of this latter group, the investigators plan to enroll 50 subjects with tympanic membrane perforation, 50 subjects with serous otitis media, 50 subjects with cholesteatoma, 50 subjects with otosclerosis, and 50 subjects with unspecified middle-ear disorders. The investigators expect that approximately 20 subjects (from all groups, normal hearing, sensorineural hearing loss, and middle-ear disorders) will be lost as screen failures or will drop from the study, and thus, the investigators will recruit an additional 20 subjects to replace these. This brings the total planned number of subjects recruited for study to 640.

Testing- All subjects will receive the same clinical and WB test battery. Each subject will be tested in one laboratory visit. Subjects will be enrolled in this study that upon otoscopic inspection of their ear canals, have no active drainage from the ears, and have ear canals free of cerumen (wax) impaction, bilaterally. Subjects who are found to have draining ears or cerumen impaction will be referred for treatment. These individuals may be enrolled in the study following successful treatment for their conditions. All subjects will have a standard pure-tone air- and bone-conduction audiogram while comfortably seated in a sound-treated booth. Standard insert earphones and a bone-conduction vibrator will be used to present the sound stimuli. Next, speech audiometry will be completed and the speech reception thresholds, uncomfortable loudness test for speech, and speech recognition scores will be obtained. Then the subjects will have a standard immittance test battery consisting of a tympanogram and acoustic reflex threshold testing. Stimuli will not exceed a level of 100 decibels hearing level (dB HL). Finally, the wideband test battery will be performed with adults seated comfortably in a sound-treated booth. A small probe with a soft rubber tip will be inserted in the subject's ear canal, and the subject will be asked to remain quiet while sounds are presented to an ear via sound sources within the probe. Responses will be measured using a miniature microphone within the probe. The tests in the wideband battery are similar to the clinical admittance battery and include ambient absorbance, absorbance tympanometry and acoustic reflex threshold. The otoacoustic emission testing is a separate measurement of inner ear function typically conducted in the clinic using different equipment.

ELIGIBILITY:
Inclusion Criteria:

Adults with normal hearing

* Veteran status
* Age between 20 and 79 years
* All puretone thresholds at 25 dB HL or lower

Adults with sensory neural hearing loss

* Veteran status
* Age between 20 and 79 years
* Average hearing thresholds between 26 and 55 dB HL

Adults with middle ear disorders

* Veteran status
* Adult between 20 and 89 years
* Diagnosis of middle ear disorder

Exclusion Criteria:

* Draining ear
* Sensory neural hearing loss greater than 55 dB HL
* Cerumen impaction of ear canal

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans will be recruited for this study who have had a hearing evaluation from the VA Audiology Service at the Portland VA Medical Center and the H. Quillen VA Medical Center. We may also recruit from approved subject registries at each study site, and from those who respond to approved fliers posted at the each site.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Patrick Feeney, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (2):
- United States (2):
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN, Mountain Home, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Hearing Adults | Adults With Sensory Neural Hearing Loss | Adults With Middle Ear Disorders
Started | 148 | 113 | 59
Completed | 108 | 83 | 54
Not Completed | 40 | 30 | 5

BASELINE CHARACTERISTICS:
Population: We consented a total of 320 participants. However, 75 were excluded because they did not meet inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hearing Adults | Adults With Sensory Neural Hearing Loss | Adults With Middle Ear Disorders | Total
Number analyzed (Participants) | 108 | 83 | 54 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 29 | 18 | 144
  >=65 years | 11 | 54 | 36 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.42 (16.12) | 66.07 (9.93) | 64.69 (12.38) | 55.78 (17.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 5 | 11 | 61
  Male | 63 | 78 | 43 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 1 | 5
  Not Hispanic or Latino | 104 | 83 | 53 | 240
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 2 | 3 | 14
  White | 90 | 79 | 51 | 220
  More than one race | 5 | 2 | 0 | 7
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 108 | 83 | 54 | 245

OUTCOME MEASURES:

1. Primary Outcome: Experimental Middle Ear Test: Ambient Wideband Absorbance
Description: Ambient Wideband Absorbance is the experimental middle ear test. Results were compared to the Secondary Outcome Measure of Clinical Peak Static Acoustic Admittance. Wideband absorbance was averaged across frequencies from 250 to 8000 Hz on a ratio scale from 0 to 1. In general, higher absorbance is indicative of a better outcome (i.e., better middle ear function).
Time Frame: Assessed at the time of enrollment during one 2.5- to 3-hour visit.
Population: Reflects total number of participants with useable data (reflects where we were in the process of developing the test battery, equipment and software issues, etc.).
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Normal Hearing Adults | Adults With Sensory Neural Hearing Loss | Adults With Middle Ear Disorders
Number analyzed (Participants) | 98 | 60 | 41
Ratio | 0.39 (0.15) | 0.38 (0.15) | 0.32 (0.21)

2. Secondary Outcome: Middle Ear Muscle Reflex Test
Description: This measure is middle ear muscle reflex thresholds in decibel (dB) sound pressure level (SPL) elicited in response to a broadband noise (BBN) activator on the standard clinical system and the experimental wideband (WB) system. The range is from 0 to 95 dB SPL with lower thresholds indicating a better outcome.
Time Frame: Assessed at the time of enrollment during one 2.5- to 3-hour visit.
Population: This outcome focused on the acoustic reflex part of the test battery which was in development longer than the other outcomes measures. The lower number of participants (in comparison to the number of Baseline Participants) included in this measure reflects the delayed addition of the reflex test to the battery, and missing data due to software or equipment issues.
Measure: Mean (Standard Deviation); unit: middle ear muscle reflex in dB SPL
Arm/Group | Normal Hearing Adults | Adults With Sensory Neural Hearing Loss | Adults With Middle Ear Disorders
Number analyzed (Participants) | 39 | 47 | 40
middle ear muscle reflex in dB SPL
  Clinical System | 85.45 (7.90) | 92.02 (3.86) | 94.36 (3.05)
  Experimental Wideband System | 69.54 (11.89) | 86.99 (7.60) | 93.27 (6.68)

3. Secondary Outcome: Wideband Otoacoustic Emission Test
Description: This measure is the difference between otoacoustic emissions and noise levels in decibels (dB) sound pressure level (SPL) elicited by a chirp averaged across frequencies from 1000 to 8000 Hertz (Hz). The normal range is ~0 to 20 dB SPL with larger values being better.
Time Frame: Assessed at the time of enrollment during one 2.5- to 3-hour visit.
Population: The lower number of participants (compared to the number of Baseline Participants) included in this measure reflects missing data due to software or equipment issues.
Measure: Mean (Standard Deviation); unit: difference level in dB SPL
Arm/Group | Normal Hearing Adults | Adults With Sensory Neural Hearing Loss | Adults With Middle Ear Disorders
Number analyzed (Participants) | 98 | 60 | 41
difference level in dB SPL | 10.29 (2.56) | 4.29 (1.06) | 3.30 (3.08)

4. Secondary Outcome: Clinical Middle Ear Test: Peak Static Acoustic Admittance
Description: Peak Static Acoustic Admittance is the standard clinical middle ear test. Results were compared to the Primary Outcome Measure of Ambient Wideband Absorbance. Peak Static Acoustic Admittance estimated from a 226-Hz tympanogram is measured on a mmho scale from 0.00 mmho to ~5.0 mmho. The normal range (i.e., normal middle ear function) is 0.3 to 1.7 mmho.
Time Frame: Assessed at the time of enrollment during one 2.5- to 3-hour visit.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: admittance in mmho
Arm/Group | Normal Hearing Adults | Adults With Sensory Neural Hearing Loss | Adults With Middle Ear Disorders
Number analyzed (Participants) | 98 | 60 | 41
admittance in mmho | 0.7 (0.24) | 0.8 (0.35) | 0.81 (0.85)

ADVERSE EVENTS:
Time Frame: Data were collected from each participant in one visit of 2.5 to 3 hours duration.
Description: Our study was deemed minimal risk by our respective Institutional Review Boards (IRBs).
Arm/Group | Normal Hearing Adults | Adults With Sensory Neural Hearing Loss | Adults With Middle Ear Disorders
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/113 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/113 | 0/59
Other Adverse Events (participants affected / at risk) | 0/148 | 0/113 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Informed Consent Form: Portland ICD (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT02019888/ICF_000.pdf
  • Informed Consent Form: Mountain Home ICD (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT02019888/ICF_001.pdf
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT02019888/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT02019888/SAP_003.pdf